CLINICAL TRIAL: NCT02051972
Title: Nanostim Study for a Leadless Cardiac Pacemaker System
Brief Title: The LEADLESS Observational Study
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: LCP005
Record Dates: First submitted 2014-01-30; First posted 2014-01-31 (Estimated); Results first posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Indications for VVI(R) Pacemaker

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Indicated for a VVI(R) pacemaker
  Interventions: Device: Implanted with a Nanostim leadless pacemaker system

INTERVENTIONS:
Device: Implanted with a Nanostim leadless pacemaker system

SUMMARY:
The objective of the study is to confirm clinical performance and safety of the Nanostim leadless cardiac pacemaker system within its intended use and according to its instructions for use.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have one of the following clinical indications: Chronic atrial fibrillation with 2 or 3° AV or bifascicular bundle branch block (BBB block) ; or Normal sinus rhythm with 2º or 3° AV or BBB block and a low level of physical activity or short expected lifespan (but at least one year); or Sinus bradycardia with infrequent pauses or unexplained syncope with EP findings; and
* Subject ≥18 years of age; and
* Subject has life expectancy of at least one year and is a suitable candidate based on overall health and well-being; and
* Subject is not enrolled in another clinical investigation with a treatment arm or that could confound the results of this study; and
* Subject is willing to comply with clinical investigation procedures and agrees to return for all required follow-up visits, tests, and exams; and
* Subject has been informed of the nature of the study, agrees to its provisions and has provided written informed consent, approved by the EC; and
* Subject is not pregnant and does not plan on getting pregnant during the course of the study.

Exclusion Criteria:

* Known pacemaker syndrome, have retrograde VA conduction or suffer a drop in arterial blood pressure with the onset of ventricular pacing; or
* Hypersensitivity to < 1 mg of dexamethasone sodium phosphate; or
* Mechanical tricuspid valve prosthesis; or
* Pre-existing pulmonary arterial (PA) hypertension (PA systolic pressure exceeds 40mmHg or RV systolic pressure (RVSP) as estimated by echo exceeds 40mmHg) or significant physiologically-impairing lung disease (has severe pulmonary disease producing frequent hospitalization for respiratory distress or requiring continuous home oxygen); or
* Pre-existing ventricular pacing or defibrillation leads; or
* Current implantation of either conventional or subcutaneous implantable cardioverter defibrillator (ICD) or cardiac resynchronization therapy (CRT); or
* Presence of implanted vena cava filter; or
* Evidence of thrombosis in one of the veins used for access during the procedure; or
* Cardiovascular or peripheral vascular surgery/intervention within 30 days of enrolment; or
* Presence of implanted leadless cardiac pacemaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who are at least 18 years old and who are indicated for a VVI(R) pacemaker
Sampling Method: Non-Probability Sample
Enrollment: 491 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2021-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Sperzel, MD, Principal Investigator — Kerckhoff Klinick GmbH, Bad Nauheim, Germany
Locations (32):
- Na Homolce Hospital, Prague, Czechia
- France (5):
  - CHRU Albert Michallon, Grenoble
  - Hopital La Timone, Marseille
  - Nouvelles cliniques Nantaises, Nantes
  - CHRU Hopital de Pontchaillou, Rennes
  - CHU Strasbourg - Hôpital de Hautepierre, Strasbourg
- Germany (9):
  - Kerckhoff-Klinik gGmbH, Bad Nauheim
  - Universitätsmedizin Berlin - Campus Benjamin Franklin, Berlin
  - Klinikum Bielefeld gGmbH Klinikum-Mitte, Bielefeld
  - Herzzentrum Dresden GmbH Universitätsklinik, Dresden
  - Asklepios Klinik St. Georg, Hamburg
  - Kath. Krankenhaus Marienhospital, Herne
  - Herzzentrum Leipzig GmbH, Leipzig
  - Deutsches Herzzentrum München des Freistaates Bayern, München
  - Kliniken Villingen-Schwenningen, Villingen-Schwenningen
- Italy (6):
  - Az. Osp. Spedali Civili di Brescia, Brescia
  - Ospedale San Raffaele, Milan
  - Ospedale Niguarda Ca'Granda, Milan
  - Centro Cardiologico Monzino, Milan
  - Policlinico San Donato, San Donato Milanese
  - Azienda Ospedaliera Bolognini, Seriate
- Netherlands (2):
  - AMC, Amsterdam
  - Isala Klinieken, Zwolle
- Spain (5):
  - Hospital Infanta Cristina, Badajoz
  - Hospital Universitario de la Paz, Madrid
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario Donostia, San Sebastián
  - Hospital do Meixoeiro, Vigo
- United Kingdom (4):
  - St. Bartholomew's Hospital, London
  - Royal Brompton Hospital, London
  - Manchester Heart Center, Manchester Royal Infirmary, Manchester
  - John Radcliffe Hospital, Oxford

REFERENCES:
- [Derived] Reddy VY, Miller MA, Knops RE, Neuzil P, Defaye P, Jung W, Doshi R, Castellani M, Strickberger A, Mead RH, Doppalapudi H, Lakkireddy D, Bennett M, Sperzel J. Retrieval of the Leadless Cardiac Pacemaker: A Multicenter Experience. Circ Arrhythm Electrophysiol. 2016 Dec;9(12):e004626. doi: 10.1161/CIRCEP.116.004626. PMID 27932427

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 491 participants were enrolled in the study but implant could be attempted in 488/491.
Groups:
- Indicated for a VVI(R) Pacemaker: Implanted with a Nanostim leadless pacemaker system
Period: Overall Study
Arm/Group | Indicated for a VVI(R) Pacemaker
Started | 488
Completed | 139
Not Completed | 349

BASELINE CHARACTERISTICS:
Population: 491 participants were enrolled in the study but implant could be attempted in 488/491. Baseline analyses include all participants enrolled
Arm/Group | Indicated for a VVI(R) Pacemaker
Number analyzed (Participants) | 491
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.8 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 182
  Male | 309
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Netherlands | 86
  Czechia | 99
  Italy | 47
  United Kingdom | 20
  France | 107
  Germany | 66
  Spain | 66
Body-Mass Index [Mean (Standard Deviation); unit: kg/m^2] — Population: Values were not taken for 2 patients, it was forgotten by the team.
  kg/m^2
    number analyzed (Participants) | 489
    (all) | 27.3 (6.6)
Weight [Mean (Standard Deviation); unit: kg] — Population: Value was not taken for 1 patient, it was forgotten by the clinical team.
  kg
    number analyzed (Participants) | 490
    (all) | 78.9 (20.9)
Height [Mean (Standard Deviation); unit: cm] — Population: Values was not taken by the clinical team
  cm
    number analyzed (Participants) | 489
    (all) | 169.8 (9.3)
LV Ejection Fraction [Mean (Standard Deviation); unit: Percentage of Left Ventricular Ejection] — Population: Ejection fraction values could not be taken in 213 participants
  Percentage of Left Ventricular Ejection
    number analyzed (Participants) | 278
    (all) | 57.8 (9.2)

OUTCOME MEASURES:

1. Primary Outcome: Complication Free-rate
Description: A complication is defined as a serious adverse device effect
Time Frame: 6 months
Population: The evaluation was completed for the first 300 subjects that completed 6 months of follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Indicated for a VVI(R) Pacemaker
Number analyzed (Participants) | 300
Participants
  Number of patients with SADEs | 16
  Number of patients free of SADEs | 284

2. Other Pre Specified Outcome: Long Term Freedom From Complications
Description: A complication is defined as a serious adverse device effect. The complication-free rate was calculated using the Kaplan-Meier method, and the 95% confidence interval was estimated using the Greenwood method.
Time Frame: 5 years
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Indicated for a VVI(R) Pacemaker
Number analyzed (Participants) | 488
percentage of patients | 55.9 [50.3 to 61.2]

3. Other Pre Specified Outcome: Long Term Freedom From Complications
Description: as for outcome 2
Time Frame: 90 days
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Indicated for a VVI(R) Pacemaker
Number analyzed (Participants) | 488
percentage of patients | 94.0 [91.5 to 95.8]

ADVERSE EVENTS:
Time Frame: The adverse event were collected over a period of 8 years
Description: The same classification criteria as clinicaltrials.gov were used for seriousness of adverse events. Adverse events are presented based on the term classified by the Sponsor. For some events, the term is the same as the organ system class.
Arm/Group | Indicated for a VVI(R) Pacemaker
All-Cause Mortality (participants affected / at risk) | 140/491
Serious Adverse Events (participants affected / at risk) | 142/491
Other Adverse Events (participants affected / at risk) | 7/491
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Indicated for a VVI(R) Pacemaker (N=491)
Decompensated HF (Cardiac disorders) | 19 (20)
Infection, Local at Access Site, Or Systemic (Skin and subcutaneous tissue disorders) | 20 (20)
Stroke (Vascular disorders) | 11 (11)
Respiratory Disease/Disorder (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Myocardial Infarction (Cardiac disorders) | 5 (5)
Cardiac Arrhythmias (Cardiac disorders) | 4 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hematoma Formation, Including, Retroperitoneal Hematoma/Hemorrhage (Vascular disorders) | 2 (2)
Excessive Bleeding (Vascular disorders) | 1 (1)
Insufficient Cardiac Output (Cardiac disorders) | 1 (1)
Pericardial Effusion (Cardiac disorders) | 1 (1)
Syncope (Cardiac disorders) | 1 (1)
General Disorders (General disorders) | 29 (29)
Neoplasms, Benign, Malignant and Unspecified Tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 24 (24)
Cardiac Disorder (Cardiac disorders) | 8 (8)
Infections and Infestations (Infections and infestations) | 4 (4)
Renal and Urinary Disorder (Renal and urinary disorders) | 4 (4)
Endocrine Disorder (Endocrine disorders) | 1 (1)
Injury, Poisoning and Procedural Complications (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Indicated for a VVI(R) Pacemaker (N=491)
Dizziness (Vascular disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Cardiac Arrhythmias (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Investigations (Product Issues) | 1 (1) — Event described as investigations involved subject exhibiting increased inflammatory markers shortly after the implant procedure. The investigator indicated that the increase may be related to the implant procedure.

LIMITATIONS AND CAVEATS:
The primary safety endpoint was met however, the supplementary endpoint of freedom from complications at 5 years was only evaluated using descriptive analyses. The enrollment goal for a powered analysis was not met since enrollments were suspended on October 28, 2016. The Nanostim LP device was not commercialized in the US and commercial sales in the EU were discontinued in 2016. The device was redesigned into the Aveir VR LP device- evaluated in the LEADLESS II Phase 2 study (NCT04559945.)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-22): https://cdn.clinicaltrials.gov/large-docs/72/NCT02051972/Prot_SAP_000.pdf